CLINICAL TRIAL: NCT03492606
Title: Specialized Pro-resolving Lipid Mediators in the Resolution of Multiple Sclerosis
Brief Title: Lipid Mediators in Multiple Sclerosis
Acronym: LipidMediators
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Mario Stampanoni Bassi, MD, Neuromed IRCCS
Other Study IDs: LipidMediators
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sampling Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple sclerosis patients
  Interventions: Procedure: Samples

INTERVENTIONS:
Procedure: Samples — lumbar puncture, blood and CSF samples, SNPs analysis

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory neurodegenerative disease associated with uncontrolled inflammation and autoimmunity and for which there is still an unmet need for new diagnostic and therapeutic options, especially for the progressive forms. Recent studies suggest that chronic inflammation can be a consequence of failure to resolve inflammation, the resolution of which is mediated by a newly discovered genus of highly potent anti-inflammatory lipids derived metabolically from omega-3 essential fatty acids and termed specialized pro-resolving lipid mediators (SPMs).

Herein, we propose to identify SPMs as leads for the control of MS pathology and progression and to propose them as novel disease-modifying treatments by assessing their ex vivo/in vitro and in vivo role in modulating the balance of effector and regulatory cells and/or the mechanisms leading to chronicity as wells as in promoting activation of anti-inflammatory and neuroprotective pathways.

DETAILED DESCRIPTION:
Uncontrolled or unresolved inflammation is associated with several widely occurring diseases such as multiple sclerosis (MS), which is the most common chronic inflammatory demyelinating disease of the central nervous system and a major cause of disability, triggered by an autoimmune response to myelin that eventually leads to progressive neurodegeneration.Although knowledge on its underlying immunopathogenesis has considerably improved and is mostly believed to be mediated by autoreactive T cells that cause oligodendrocyte death and axonal damage, resulting in demyelination, synaptic alteration, and neuronal loss, there is still an unmet need for new diagnostic and therapeutic options, especially for the progressive forms of MS for which no drugs are still available. In recent years, previously unrecognized metabolites, termed specialized pro-resolving lipid mediators (SPMs), temporally and spatially synthesized from omega-3 polyunsaturated fatty acids, were identified and have emerged as biomarkers and potent mediators that control the magnitude and extent of inflammatory events by activating local resolution programs. Despite emerging data suggest that SPMs might control chronic inflammation, research on these mediators on MS is still absent. Thus, a detailed investigation is needed to identify SPMs as modulators of inflammation and disease progression in MS, which might lead to the development of new disease-modifying treatments.

Hypothesis and Significance:

Our hypothesis is that the underlying mechanism of chronic inflammation in MS could be the failure of activating pro-resolving mechanisms, involving the newly discovered omega-3 essential fatty acids-derived mediators of resolution of inflammation: resolvins, maresins, and protectins. Endogenous mechanisms that curtail excessive inflammation and promptits timely resolution are of considerable interest; our findings that these SPMs (recently identified also in human lymphoidorgans, where most naïve-to-effector T cell differentiation occurs) exert a non-cytotoxic regulatory role on cells central inautoimmunity, acting on the balance between pathogenic Th1/Th17 and tolerogenic Treg cells - typically altered in MS -represents a promising beginning for a new avenue of research for MS. The elucidation of these mechanisms operating invivo to keep acute inflammation within physiologic boundaries as well as to stimulate resolution and prevent chronicinflammation is particularly significant and offers a novel opportunity to manage MS.

Preliminary Data:

Thanks to an ongoing collaboration with Prof. Serhan from Harvard Medical School (the father and inventor of SPMs) we have demonstrated for the first time that specific SPMs modulate adaptive immune responses in human peripheral blood T cells. These SPMs strongly reduce cytokine production from activated T cells, prevent naïve CD4 T-cell differentiation into Th1 and Th17 and enhance the de novo generation and function of Foxp3+ regulatory T (Tregs) cells. These results are supported in vivo in a mouse model deficient elongase 2 (Elovl2-/-), the key enzyme for DHA synthesis (the precursor of resolvins and maresins). These findings suggest that SPMs might act on the balance between pathogenic Th1/Th17 and tolerogenic Treg cells and provide a new evidence for SPM-based therapeutic approaches to modulate T-cell mediated chronic inflammatory and autoimmune diseases.

Specific Aims:

Characterization of the resolution code of inflammation in MS patientsInvestigation of SPMs potential in modulating ex vivo/in vitro T cells in MS patientsExploitation of the therapeutic potential of SPMs in animal models of MS

ELIGIBILITY:
Inclusion Criteria:

Inclusion in the study is foreseen for sex subjects, ideally in a ratio of 1: 2.5 in favor of the female (according to the incidence of the disease), aged between 18 and 60 years, affected by the recurrent form - Multiple sclerosis emitter with EDSS between 1 and 3. Blood sampling will be performed at least one month after the last cortisone treatment. Taking into account that 20% of the enrolled patients could have a variability in the cell count of the monocytes to be purified, the number of the sample up to 24 is better than 20%.

Exclusion Criteria:

Subjects who have at least one of the following characteristics will not be included in the study:

1. subjects with CNS or autoimmune diseases
2. subjects affected by RR-MS in immunomodulatory treatment
3. subjects with RR-MS with monocytosis, infections or fever

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 20 recurrent-remitting patients (RR-MS) and 10 primary-progressive patients (P-MS), according to the MacDonald or Poser method, without any type of treatment and 15 healthy donors of the same age and with no previous history of neurological diseases. Blood samples will be recruited at the IRCCS INM Neuromed, under the supervision of dr. Fabio Buttari who will make the diagnosis. The diagnosis of MS will be performed according to the criteria of MacDonald or Poser. On this occasion, the patient will be offered participation in the study, giving informed consent and explaining in non-technical language, what the research consists of, which parameters will be evaluated and for what purpose. Once consent is obtained from the patients, venous samples will be taken (15 mL).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
SPMs in plasma | 2021
  levels of the different members of the family of SPMs in plasma
T cells | 2021
  analysis of T cells functions
EAE | 2021
  we will treat acute EAE mice (n=8 per each experimental group) at the peak of the disease (day 16-19) with those SPMs that will result to be the most efficacious in modulating pathogenic T-cell responses

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No